CLINICAL TRIAL: NCT04702893
Title: Prospective Observational Investigation of Possible Correlations Between Change in FVC and Change in Cough or Dyspnea Scores Using the Living With Pulmonary Fibrosis Questionnaire (L-PF) Between Baseline and After Approximately 52 Weeks of Nintedanib Treatment in Patients Suffering From Chronic Fibrosing ILD With a Progressive Phenotype
Brief Title: INREAL - Nintedanib for Changes in Dyspnea and Cough in Patients Suffering From Chronic Fibrosing Interstitial Lung Disease (ILD) With a Progressive Phenotype in Everyday Clinical Practice: a Real-world Evaluation
Acronym: INREAL
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0449
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nintedanib-treated patients: Patients diagnosed with chronic fibrosing interstitial lung disease (ILD) with a progressive phenotype (excluding idiopathic pulmonary fibrosis (IPF)), who did not receive previous antifibrotic treatment, received 150 milligrams (mg) of nintedanib twice daily, administered 12 hours apart, according to the approved label, for approximately 52 weeks. Participants who did not tolerate 150 mg of nintedanib switched to 100 mg twice daily.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — 150 or 100 milligrams (mg) of nintedanib, when 150 mg is not tolerated, twice daily, administered 12 hours apart, according to the approved label.
  Other Names: Ofev®

SUMMARY:
The primary objective of this observational study is to investigate the correlation between changes from baseline at 52 weeks in forced vital capacity (FVC) and changes from baseline at 52 weeks in dyspnea score points or cough score points as measured with the pulmonary fibrosis questionnaire (L-PF) questionnaire over 52 weeks of nintedanib treatment in patients suffering from chronic fibrosing interstitial lung disease (ILD) with a progressive phenotype (excluding idiopathic pulmonary fibrosis (IPF)).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years at Visit 1
* Subjects must be contractually capable and mentally able to understand and follow the instructions of the study personnel
* Physician's diagnosis of chronic fibrosing interstitial lung disease (ILD) with a progressive phenotype, except idiopathic pulmonary fibrosis (IPF)
* Treatment with nintedanib in INREAL will be the first and only prescription of any antifibrotic treatment for each individual patient within this observational study after a physician's decision being made for this treatment option earlier
* Outpatients not currently hospitalized with a life expectancy > 12 months per investigator's assessment
* Written informed consent prior to study participation
* Current forced vital capacity (FVC) measurement (taken within the last 3 months) available in the patient file
* Women of childbearing potential must take appropriate precautions against getting pregnant during the intake of nintedanib

Exclusion Criteria:

* Patients with contraindications according to Summary of Product Characteristics (SmPC)
* Prior use of any antifibrotic treatment
* Lack of informed consent
* Pregnant or lactating females
* Any physician diagnosed exacerbation of ILD in the patient's history file, irrespective of time since event
* Current diagnosis of lung cancer
* Respiratory failure (pH < 7,35 and/ or respiratory rate > 30/min) in the patient's history
* Participation in a parallel interventional clinical trial
* Patients being spouse or lateral relatives to the second degree or economically dependent from the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this NIS, data on the effect of nintedanib in chronic fibrosing ILD with progressive phenotype in about 100 patients will be collected in routine clinical practice by ca. 20 specialists, experienced in treating ILD patients, (e. g. pulmonologists and rheumatologists) throughout Germany.
  Patients to be recruited within this study have to have a physician diagnosed chronic fibrosing interstitial lung disease (ILD) with a progressive phenotype (except idiopathic pulmonary fibrosis (IPF)), for which nintedanib is an indicated treatment.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Marseille, +4961327714188, Study Chair — andrea.marseille@boehringer-ingelheim.com
Locations (21):
- Germany (21):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Pneumologische Praxis Dr. Löh, Bad Homburg
  - ACURA Kliniken Rheinland-Pfalz, Bad Kreuznach
  - Vivantes Klinikum Neukölln, Berlin
  - Klinikum Braunschweig, Braunschweig
  - Klinikum Chemnitz, Chemnitz
  - Kliniken der Stadt Köln, Cologne
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Universitätsklinikum Erlangen, Erlangen
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Praxis Dr. med. Claus Keller, Frankfurt
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg Thoraxklinik Heidelberg Zentrum für interstitielle und seltene Lungenerkrankungen, Heidelberg
  - Lungenklinik Hemer in der Trägerschaft der Deutschen Gemeinschafts-Diakonieverband GmbH, Hemer
  - Rheumazentrum Herne, Herne
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Lippe, Lemgo
  - Johannes Wesling Klinikum Minden der Mühlenkreiskliniken AöR, Minden
  - Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen
  - Petrus-Krankenhaus, Wuppertal

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single-arm, open-label observational cohort study investigating the effect of nintedanib on patient-reported outcomes (PROs) like dyspnea and cough in chronic interstitial lung disease (ILD) patients (excluding idiopathic pulmonary fibrosis (IPF)) over 52 weeks.
Pre-assignment Details: Only patients that met all inclusion and none of the exclusion criteria were included.
Period: Overall Study
Arm/Group | Nintedanib-treated Patients
Started | 108
Treated | 102
Completed | 71
Not Completed | 37
Not completed — Other reasons than listed | 11
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 7
Not completed — Death | 10
Not completed — Not treated | 6

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients with signed informed consent who received at least one dose of nintedanib.
Arm/Group | Nintedanib-treated Patients
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.47 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Forced vital capacity (FVC) [% predicted] [Mean (Standard Deviation); unit: Percentage] — Population: Only TS patients without missing baseline data were included.
  Percentage
    number analyzed (Participants) | 98
    (all) | 65.18 (18.86)
Living with pulmonary fibrosis questionnaire (L-PF) dyspnea symptom score [Mean (Standard Deviation); unit: Units on a scale] — The L-PF includes a dyspnea symptom module with 12 items to evaluate the severity of dyspnea symptoms. Each item is scored on a scale of 0 to 5, with higher scores indicating more severe symptoms. The total dyspnea symptom score was calculated using the formula: (sum of each individual score/total score possible)*100, ranging from 0 to 100, where the higher the score, the more severe the dyspnea. Population: Only TS patients without missing baseline data were included.
  Units on a scale
    number analyzed (Participants) | 101
    (all) | 24.71 (18.56)
Living with pulmonary fibrosis questionnaire (L-PF) cough symptom score [Mean (Standard Deviation); unit: Units on a scale] — The L-PF includes a cough symptom module with 6 items to evaluate the severity of cough symptoms. Each item is scored on a scale of 0 to 4, with higher the scores indicating more severe symptoms. The total cough symptom score was calculated using the formula: (sum of each individual score/24)*100, ranging from 0 to 100, where the higher the score, the more severe the cough. Population: Only TS patients without missing baseline data were included.
  Units on a scale
    number analyzed (Participants) | 101
    (all) | 37.46 (25.67)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Change From Baseline to Week 52 in Forced Vital Capacity (FVC) [% Predicted] and Change From Baseline to Week 52 in Dyspnea Symptom Score
Description: The correlation between the change from baseline to week 52 (week 52 - baseline) in forced vital capacity (FVC) [% predicted] and change from baseline to week 52 (week 52 - baseline) in dyspnea symptom score was calculated using the Pearson's coefficient of correlation. The forced vital capacity measures the amount of air that can be forcefully exhaled from the lungs after a maximum inhalation. The dyspnea symptom score was measured using the living with pulmonary fibrosis questionnaire (L-PF). The L-PF contained a dyspnea symptom module with 12 items to assess the severity of shortness of breath, where the higher the score, the greater the impairment. The coefficient of correlation ranges from -1 to 1, indicating a negative association between the variables the closer it is to -1 and a positive association the closer it is to 1.
Time Frame: At baseline and at week 52±6.
Population: Treated set (TS): All patients with signed informed consent who received at least one dose of nintedanib. Patients with missing data were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: Pearson's coefficient of correlation
Arm/Group | Nintedanib-treated Patients
Number analyzed (Participants) | 38
Pearson's coefficient of correlation | -0.2576 [-0.5333 to 0.0677]
Statistical Analysis 1: Comparison: Nintedanib-treated Patients; Test type: Other — No formal hypotheses were tested; p = 0.1185, Z-test of correlation

2. Primary Outcome: Correlation Between Change From Baseline to Week 52 in Forced Vital Capacity (FVC) [% Predicted] and Change From Baseline to Week 52 in Cough Symptom Score
Description: The correlation between the change from baseline to week 52 (week 52 - baseline) in forced vital capacity (FVC) [% predicted] and change from baseline to week 52 (week 52 - baseline) in cough symptom score was calculated using the Pearson's coefficient of correlation. The forced vital capacity measures the amount of air that can be forcefully exhaled from the lungs after a maximum inhalation. The cough symptom score was measured using the living with pulmonary fibrosis questionnaire (L-PF). The L-PF contained a cough symptom module with 6 items to assess the severity of cough symptoms, where the higher the score, the more severe the cough. The coefficient of correlation ranges from -1 to 1, indicating a negative association between the variables the closer it is to -1 and a positive association the closer it is to 1.
Time Frame: At baseline and at week 52±6.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Pearson's coefficient of correlation
Arm/Group | Nintedanib-treated Patients
Number analyzed (Participants) | 38
Pearson's coefficient of correlation | -0.1093 [-0.4145 to 0.2180]
Statistical Analysis 1: Comparison: Nintedanib-treated Patients; Test type: Other — No formal hypotheses were tested; p = 0.5135, Z-test of correlation

3. Secondary Outcome: Correlation Between Change From Baseline to Week 52 in Forced Vital Capacity (FVC) [mL] and Change From Baseline to Week 52 in Dyspnea Symptom Score
Description: The correlation between the change from baseline to week 52 (week 52 - baseline) in forced vital capacity (FVC) [mL] and change from baseline to week 52 (week 52 - baseline) in dyspnea symptom score was calculated using the Pearson's coefficient of correlation. The forced vital capacity measures the amount of air that can be forcefully exhaled from the lungs after a maximum inhalation. The dyspnea symptom score was measured using the living with pulmonary fibrosis questionnaire (L-PF). The L-PF contained a dyspnea symptom module with 12 items to assess the severity of shortness of breath, where the higher the score, the greater the impairment. The coefficient of correlation ranges from -1 to 1, indicating a negative association between the variables the closer it is to -1 and a positive association the closer it is to 1.
Time Frame: At baseline and at week 52±6.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Pearson's coefficient of correlation
Arm/Group | Nintedanib-treated Patients
Number analyzed (Participants) | 38
Pearson's coefficient of correlation | -0.2909 [-0.5587 to 0.0317]
Statistical Analysis 1: Comparison: Nintedanib-treated Patients; Test type: Other — No formal hypotheses were tested; p = 0.0764, Z-test of correlation

4. Secondary Outcome: Correlation Between Change From Baseline to Week 52 in Forced Vital Capacity (FVC) [mL] and Change From Baseline to Week 52 in Cough Symptom Score
Description: The correlation between the change from baseline to week 52 (week 52 - baseline) in forced vital capacity (FVC) [mL] and change from baseline to week 52 (week 52 - baseline) in cough symptom score was calculated using the Pearson's coefficient of correlation. The forced vital capacity measures the amount of air that can be forcefully exhaled from the lungs after a maximum inhalation. The cough symptom score was measured using the living with pulmonary fibrosis questionnaire (L-PF). The L-PF contained a cough symptom module with 6 items to assess the severity of cough symptoms, where the higher the score, the more severe the cough. The coefficient of correlation ranges from -1 to 1, indicating a negative association between the variables the closer it is to -1 and a positive association the closer it is to 1.
Time Frame: At baseline and at week 52±6.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Pearson's coefficient of correlation
Arm/Group | Nintedanib-treated Patients
Number analyzed (Participants) | 38
Pearson's coefficient of correlation | -0.1566 [-0.4536 to 0.1717]
Statistical Analysis 1: Comparison: Nintedanib-treated Patients; Test type: Other — No formal hypotheses were tested; p = 0.3478, Z-test of correlation

5. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis Questionnaire (L-PF) Cough Symptom Score [Points] at Week 52
Description: This outcome measured the absolute change from baseline to week 52 in the cough symptom score, assessed by the living with pulmonary fibrosis questionnaire (L-PF). The L-PF includes a cough symptom module with 6 items to evaluate the severity of cough symptoms. Each item is scored on a scale of 0 to 4, with higher scores indicating more severe symptoms. The total cough symptom score was calculated using the formula: (sum of each individual score/24)*100, ranging from 0 to 100, where the higher the score, the more severe the cough. Results were calculated as [Week 52] - [Baseline].
  The analysis was performed using a mixed model for repeated measures (MMRM) with fixed independent effects for baseline value, visit, and baseline-by-visit interaction, and a random effect for each patient. Within-patient errors were represented using an unstructured variance-covariance structure.
Time Frame: MMRM included measurements at week 13±6, week 26±6, week 39±6 and week 52±6. Change from baseline values at week 52±6 is reported.
Population: Treated set (TS): All patients with signed informed consent who received at least one dose of nintedanib. Only patients with at least one post baseline value and baseline value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Nintedanib-treated Patients
Number analyzed (Participants) | 91
Units on a scale | 3.86 (3.28)

6. Secondary Outcome: Absolute Change From Baseline in Living With Pulmonary Fibrosis Questionnaire (L-PF) Dyspnea Symptom Score [Points] at Week 52
Description: This outcome measured the absolute change from baseline to week 52 in the dyspnea symptom score, assessed by the living with pulmonary fibrosis questionnaire (L-PF). The L-PF includes a dyspnea symptom module with 12 items to evaluate the severity of dyspnea symptoms. Each item is scored on a scale of 0 to 5, with higher scores indicating more severe symptoms. The total dyspnea symptom score was calculated using the formula: (sum of each individual score/total score possible)*100, ranging from 0 to 100, where the higher the score, the more severe the dyspnea. Results were calculated as [Week 52] - [Baseline].
  The analysis was performed using a mixed model for repeated measures (MMRM) with fixed independent effects for baseline value, visit, and baseline-by-visit interaction, and a random effect for each patient. Within-patient errors were represented using an unstructured variance-covariance structure.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Nintedanib-treated Patients
Number analyzed (Participants) | 91
Units on a scale | 6.26 (2.35)

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality: From first nintedanib administration to 52±6 weeks thereafter plus 28 days of residual effect period. Up to 62 weeks.
Description: Treated set (TS): All patients with signed informed consent who received at least one dose of nintedanib.
Arm/Group | Nintedanib-treated Patients
All-Cause Mortality (participants affected / at risk) | 10/102
Serious Adverse Events (participants affected / at risk) | 16/102
Other Adverse Events (participants affected / at risk) | 45/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib-treated Patients (N=102)
Myocardial infarction (Cardiac disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 1
Sudden death (General disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Nasal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Inflammatory marker increased (Investigations) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prerenal failure (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib-treated Patients (N=102)
Diarrhoea (Gastrointestinal disorders) | 42
Nausea (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT04702893/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04702893/SAP_001.pdf